CLINICAL TRIAL: NCT03535285
Title: Evaluation of Periodontal Ligament Distraction Using a Modified Surgical Technique for Retraction of Maxillary Canines in Adult Patients (Split-mouth Randomized Clinical Trial)
Brief Title: Evaluation of Periodontal Ligament Distraction Using a Modified Surgical Technique for Retraction of Maxillary Canines
Acronym: [PLD]
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Monaser Mobarak, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11111
Record Dates: First submitted 2018-05-10; First posted 2018-05-24 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Orthodontic Appliance Complication
Keywords: periodontal ligament; dentoalveolar; distraction; orthodontic

STUDY DESIGN:
Intervention Model Description: Split-mouth
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical modification side (Experimental): Periodontal ligament distraction without the oblique cuts but with apical horizontal cut
  Interventions: Procedure: Periodontal ligament distraction
- Conventional surgery (Active Comparator): Periodontal ligament distraction
  Interventions: Procedure: Periodontal ligament distraction

INTERVENTIONS:
Procedure: Periodontal ligament distraction — decrease the bony resistant during canine retration
  Other Names: Acceleration of canine retraction

SUMMARY:
Surgical modification technique try to get bodily movement during upper canine retraction.

DETAILED DESCRIPTION:
I- Original surgical technique (Liou and Huang technique, 1998) :

On the conventional surgical side, (the control side), the intersepital bone was undermined by two vertical cuts on the mesio-buccal and mesio-palatal line angles of the first premolar socket. They were connected at the base of the socket by an oblique cut. The surgical round bur was held parallel to the long axis of the canine and moved buccolingually, while shaving the interseptal bone buccolingual (back-and-forth) shaving movements were reduced the thickness of the interseptal bone by approximately 1 mm

II- Modified surgical technique:

In the surgical modification side, (the experimental side), intra-alveolar mesio-buccal and mesio-palatal cuts and interseptal bone shaving were done by surgical round bur and copious irrigation, without the oblique cut since it was done blindly in the original surgical technique. A buccal semilunar flap was opened on the apical area of canine-premolar region. The surgical pin helped also in location of the point of initial drilling of the apical horizontal cut from buccal approach, when the surgical pin's socket arm rested on the depth of the socket, the vestibular arm marked the point of access. It also estimated mesiodeistal extension of the apical horizontal cut. The apical horizontal cut was started from the socket apex to half way of the interseptal bone mesiodistally as an extension and for the depth, Mallet and Chisel were used from the cortical bone to reach the mesio-palatal cut. The flap was sutured. This surgical modification step provided more predictability and safer surgery than the blind oblique cut in the original surgical technique.

ELIGIBILITY:
Inclusion Criteria:

1. Orthodontic patients needed extraction of upper first premolars, with age range from 18 - 25 years old.
2. All patients were medically free. (See Appendix II)
3. No previous orthodontic treatment.
4. Adequate oral hygiene and periodontally healthy teeth.
5. The canines were almost leveled and aligned.
6. Maximum anchorage requirements.
7. Healthy canines; no deep carious lesions, no endodontic lesions, no root canal treatment, nor internal or external root resorption.
8. All patients were informed of the procedure and signed the consents.

Exclusion Criteria:

Exclusion Criteria

Subjects were excluded from the study when:

1. They failed to keep several consecutive appointments.
2. Oral hygiene was subjectively judged as deteriorating during the preliminary stages of patient preparation.
3. Compliance with the instructions provided was inadequate.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Tipping of the canines | 3-4 weeks
  1. Periapical radiograph using Parallel technique (X-ray sensor , X-ray sensor holder & Potable dental x-ray unit
  2. Panoramic radiograph .
Rate of canines retraction | 3-4 weeks
  Digital models using 3shape scanner and Ortho-Analyzer software
Rotation of the canines | 3-4 weeks
  Digital models using 3shape scanner and Ortho-Analyzer software

SECONDARY OUTCOMES:
Amount of anchorage loss | 3-4 weeks
  Digital models using 3shape scanner and Ortho-Analyzer software
Tipping of the molars | 3-4 weeks
  1. Periapical radiograph using Parallel technique (X-ray sensor , X-ray sensor holder & Potable dental x-ray unit
  2. Panoramic radiograph.
The apical root resorption scores | 3-4 weeks
  Periapical radiograph using Parallel technique (x-ray sensor, X-ray sensor holder & Potable dental x-ray unit
Pulp Vitality | 3-4 weeks
  Cold application (Ethyl Chloride)
Gingival index | 3-4 weeks
  Periodontal probe
Periodontal index | 3-4 weeks
  Periodontal probe
Pain | 3-4 weeks
  Numeric rating scale (NRS) for pain

CONTACTS AND LOCATIONS:
Overall Officials: Monaser M Elashik, Master, Principal Investigator — Cairo University
Locations (1):
- Cairo University - Orthodontic department, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Liou EJ, Huang CS. Rapid canine retraction through distraction of the periodontal ligament. Am J Orthod Dentofacial Orthop. 1998 Oct;114(4):372-82. doi: 10.1016/s0889-5406(98)70181-7. PMID 9790320
- See also: periodontal ligament distraction — https://www.ncbi.nlm.nih.gov/pubmed/?term=Liou+and+Huang+%5Bauthor%5D++periodontal+ligament+distracrion